CLINICAL TRIAL: NCT03196856
Title: Effects of Greek Yogurt and Exercise on Muscle Size, Body Composition and Bone Health in Untrained, University-aged Males
Brief Title: Brock Exercise And Supplement Trials
Acronym: BEAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Andrea Josse, Assistant Professor, Brock University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB16-295
Record Dates: First submitted 2017-06-14; First posted 2017-06-23 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Untrained; Healthy
Keywords: Greek Yogurt; Muscle Size; Bone Health; Body Composition; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Masking Description: Participants will be randomly selected to the yogurt group or a placebo group. Although participants within the yogurt group will be aware that they are consuming yogurt, the placebo group will not be aware of the contents of the placebo supplement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yogurt Group (Experimental): Group will be consuming 200g of Greek Yogurt (Plain, 0%) 3 times daily for 12 weeks
  Interventions: Behavioral: Resistance and Plyometric Exercise; Dietary Supplement: Greek Yogurt (0% Plain)
- Study Designed Supplement Group (Placebo Comparator): Group will consume an isoenergetic, protein void, maltodextrin-based placebo supplement during the same time points for 12 weeks as well. The Placebo contain maltodextrin and pudding powder to mimic the consistency of Greek yogurt.
  Interventions: Behavioral: Resistance and Plyometric Exercise; Dietary Supplement: Placebo - Study Designed Supplement

INTERVENTIONS:
Behavioral: Resistance and Plyometric Exercise — 12 weeks of Resistance (twice weekly) and Plyometric (once weekly) training
Dietary Supplement: Greek Yogurt (0% Plain) — 200g 3x/day for 12 weeks.
  Arms: Yogurt Group
Dietary Supplement: Placebo - Study Designed Supplement — Iso-energetic to yogurt. 3x/day for 12 weeks.
  Arms: Study Designed Supplement Group

SUMMARY:
This study will analyze the effects of Greek yogurt consumption and an 12 week exercise intervention on muscle size, body composition and bone health in untrained, university-aged males.

DETAILED DESCRIPTION:
Introduction: Previous research has shown the effectiveness of dairy milk and whey protein on increasing muscle size, optimizing body composition and increasing strength in adult males. However, evidence on the use of high protein/Greek yogurt on muscle size, body composition and bone health is limited in this population. Yogurt contains similar muscle and bone supporting nutrients as milk, yet it offers a host of additional benefits including; increased satiety, probiotic cultures, greater stability, increased variety, more affordable and versatile features such as acting as a vehicle for consumption of other healthful foods. The proposed research will investigate the use of Greek yogurt as an effective post-exercise food to promote healthy body composition and bone health changes in young adult males.

Design: Parallel, randomized controlled trial.

Participants: 30 (n=15 YOG, n=15 PLA) healthy, untrained university-aged males.

Methods: Subjects will undergo a 12-week resistance and plyometric training program (exercising 3 days/week). The YOG group will consume a 200g dose (pro= 20g, carbs= 8 grams, ~110 kcals) of plain 0% Greek yogurt, while the PLA group will consume an isoenergetic, protein-void beverage comprised mainly of maltodextrin (pro= 0g, carbs= 26g, ~110 kcals). Each group will consume 3 doses per day (immediately and 1 hour post-exercise, and bedtime). Markers of bone health (CTx and P1NP) will be taken at baseline, 1 week and 12 weeks to determine acute and total changes. Muscle size, body composition, strength, vertical jump height and nutritional diaries will be measured pre and post intervention and habitual diet maintenance will be encouraged throughout the intervention.

Anticipated Results: It is hypothesized that each group will undergo positive changes in the aforementioned measures, however due to the increase in protein and calcium consumption, the yogurt group is predicted to have significantly greater increases in these variables than the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-25 years
* Normal BMI (18.5-24.9) kg/m2
* Have not participated in a resistance training program (of resistance exercise at least 2x/week or more) in the last 6 months
* Healthy and not taking any medication affecting muscle or bone
* Not supplementing with vitamins/ minerals or protein
* Speak and understand English
* No dairy allergy or lactose intolerance

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Muscular Strength | Change from Baseline to 12 weeks
  1 Repetition Maximum of bench press, seated row, quad extension and hamstring curl
Muscle Size | Change from Baseline to 12 weeks
  Muscle Size determined by ultrasound at various sites.
Body Composition | Change from Baseline to 12 weeks
  Body Fat % measured via BodPod and BodyMetrix

SECONDARY OUTCOMES:
Bone cell activity | Change from Baseline to 12 weeks
  Bone markers measured in serum.
Vertical Jump Height | Change from Baseline to 12 weeks
  measured via chalk-on-wall technique

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Josse, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bridge A, Brown J, Snider H, Nasato M, Ward WE, Roy BD, Josse AR. Greek Yogurt and 12 Weeks of Exercise Training on Strength, Muscle Thickness and Body Composition in Lean, Untrained, University-Aged Males. Front Nutr. 2019 Apr 30;6:55. doi: 10.3389/fnut.2019.00055. eCollection 2019. PMID 31114790
- See also: Published Manuscript — https://www.frontiersin.org/articles/10.3389/fnut.2019.00055/full